CLINICAL TRIAL: NCT01929070
Title: A Pilot Study to Evaluate the Pharmacokinetics of Omega-3 Between Rosuvastatin and Omega-3 Coadministration and HCP1007 in Healthy Male Volunteers
Brief Title: A Pilot Study to Evaluate the Pharmacokinetics of Omega-3 Between Rosuvastatin and Omega-3 Coadministration and HCP1007
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROMA-103P
Record Dates: First submitted 2013-03-14; First posted 2013-08-27 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: HCP1007; Rosuvastatin; Omega-3
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): * R1: Coadministration of Crestor 5mg 4tab and Omacor capsupe 1g 4cap in the fasting state
  * R2: Coadministration of Crestor 5mg 4tab and Omacor capsupe 1g 4cap on the high-fat diet
  * T1: Single-dose of HCP1007 1g/5mg 4 cap in the fasting state
  * T2: Single-dose of HCP1007 1g/5mg 4 cap on the high-fat diet
  R1 -> T2 -> R2 -> T1
  Interventions: Drug: HCP1007; Drug: Omarco and Crestor
- Group 2 (Experimental): R2 -> R1 -> T1 -> T2
  Interventions: Drug: HCP1007; Drug: Omarco and Crestor
- Group 3 (Experimental): T1 -> R2 -> T2 -> R1
  Interventions: Drug: HCP1007; Drug: Omarco and Crestor
- Group 4 (Experimental): T2 -> T1 -> R1 -> R2
  Interventions: Drug: HCP1007; Drug: Omarco and Crestor

INTERVENTIONS:
Drug: HCP1007
Drug: Omarco and Crestor

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of omega-3 between rosuvastatin and omega-3 coadministration and HCP1007 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult male aged 20 to 55 years
* A body mass index between 19 and 27 kg/m2

Exclusion Criteria:

* History of hepatobiliary, renal, gastrointestinal, respiratory, musculoskeletal, endocrinal, hemato-oncologic or cardiovascular disease
* SBP < 90 or ≥ 150 mmHg, DBP < 60 or ≥90 mmHg
* Use of herbal medicine within 30 days, prescriptive medicine within 14 days, or over-the-counter drug within 7 days
* Heavy alcohol consumption (140 g/day)

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cmax_adj of DHA and EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h (on the high-fat diet only)
AUClast_adj of DHA and EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h (on the high-fat diet only)

SECONDARY OUTCOMES:
Cmax of DHA, EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h(only on the high fat diet)
AUClast of DHA, EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h(only on the high fat diet)
AUClast of DHA and EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h(only on the high fat diet)
tmax of DHA and EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h(only on the high fat diet)
t1/2 of DHA and EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h(only on the high fat diet)
AUCinf of DHA and EPA | -24, -22, -20, -19, -18, -16, -14, -12, 0 (predose), 2, 4, 5, 6, 8, 10, 12, 24, 48 h, 72 h(only on the high fat diet)

CONTACTS AND LOCATIONS:
Overall Officials: JaeWook Ko, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea